CLINICAL TRIAL: NCT06915077
Title: Personalized Treatment for Obstructive Sleep Apnea: Beyond CPAP
Brief Title: Personalised Treatment for OSA
Status: Enrolling by invitation | Type: Observational
Sponsor: University Hospital, Antwerp (Other)
Responsible Party: Sponsor
Other Study IDs: EDGE 3513
Record Dates: First submitted 2025-02-11; First posted 2025-04-08 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-01

CONDITIONS: Sleep Apnea Syndrome (OSAS); Sleep Apnea Syndrome; Sleep Apnea Syndrome, Obstructive; Sleep Apnea/Hypopnea Syndrome; Sleep Apnea
MeSH Terms: conditions — Sleep Apnea Syndromes; Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Obstructive sleep apnea (OSA) is a sleep disorder characterized by repetitive episodes of partial or complete obstruction of the upper airway during sleep. Continuous positive airway pressure (CPAP) is a method used as a first-line treatment for obstructive sleep apnea (OSA). However, intolerance and resistance to CPAP can limit its long-term effectiveness. Alternative treatments are available, such as Mandibular Advancement Devices (MADs), positional therapy, upper airway surgery, and maxillomandibular osteotomy. However, often less efficient in reducing the apnea-hypopnea index, the higher tolerance of and compliance to alternative treatment has resulted in the adequate treatment of OSA in CPAP-intolerant patients. This paper describes the protocol of a prospective single-center cohort study including adult patients with moderate to severe OSA (15 events/h ≤ apnea-hypopnea index (AHI) < 65 events/h) that failed to comply with CPAP therapy. Selected patients will be invited to the clinic to explore alternative treatment options where DISE will be a first step in further identifying upper airway collapse during sleep. By exploring alternative treatment options in CPAP-intolerant patients and systematically documenting their treatment paths, an algorithm can be defined to better guide patients towards personalized treatment for OSA. The follow-up is aimed at 5 years with an inclusion of 170 patients per year, including a drop-out rate of 15%. By leveraging a real-world database, this study aims to bridge the gap between research and clinical practice, facilitating the development of evidence-based guidelines and personalized treatment algorithms for CPAP-intolerant patients.

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) is a sleep disorder characterized by repetitive episodes of partial or complete obstruction of the upper airway during sleep, leading to reduced or completely stopped airflow despite ongoing respiratory efforts. This results in disrupted sleep and intermittent hypoxia. This disorder is estimated to affect 17% of middle-aged women and 34% of middle-aged men [1]. Loud snoring, a precursor of OSA, is even more prevalent and is estimated to affect 40-60% of adult people [2]. OSA does not only cause symptoms such as excessive daytime sleepiness, loud snoring, and interrupted breathing during sleep. OSA can have significant health implications, including increased risk of hypertension, cardiovascular disease, and impaired cognitive function in the long term, as shown in several scientific studies [3,4,5]. Although 80% of patients remain undiagnosed, increasing awareness is seen over the last years [6].

OSA is diagnosed with an overnight polysomnography in a hospital setting or at home, in patients who are clinically and anamnestically suspected of OSA. Symptoms are habitual snoring, choking or gasping during sleep, excessive daytime sleepiness, inattention, and poor recall. Severity of OSA is measured using the apnea-hypopnea index (AHI), the number of apneas and hypopneas per hour of sleep. The diagnosis is confirmed if the AHI is at least five events per hour of sleep. Severity based on AHI is defined as follows: mild OSA (5 < AHI ≤ 15/h), moderate OSA (15 < AHI < 30/h) and severe OSA (AHI ≥ 30/h) [7].

Continuous positive airway pressure (CPAP) is a method used as first-line treatment for OSA. CPAP therapy significantly reduces disease severity, sleepiness, blood pressure, and sleepiness-related traffic accident occurrence, as well as improves the sleep-related quality of life in adults with sleep apnea [8].

However, intolerance and resistance to CPAP can limit its long-term effectiveness. Various factors contribute to CPAP intolerance, including mask discomfort, claustrophobia, nasal congestion, air leaks, pressure intolerance, and difficulty adjusting to the therapy [9]. Compliance failure is reported to be different in various countries. A recent nation-wide French database study showed that almost half of patients on CPAP therapy terminate the CPAP treatment after three years [10]. Therefore, alternative treatment options in CPAP-intolerant or non-compliant patients have gain increased interest and importance in daily practice, leading us towards a more personalized way of treatment.

Alternative treatments for OSA include Mandibular Advancement Devices (MADs), positional therapy, upper airway surgery, and maxillomandibular osteotomy [11,12,13,14]. MAD therapy has emerged as a second-line conservative non-invasive treatment method for the management of mild to moderate OSA, and lately even for severe OSA patients. MAD therapy consists of a titratable duo-block with separate upper and lower parts that are dynamically interconnected. This allows for a gradual protrusion of the lower jaw until the optimal position is reached. As such, patients can optimize the ideal position that allows symptoms (such as snoring and tiredness) to disappear and to tolerate protrusion as well. MAD therapy functions on increasing the upper airway volume, mainly the widening of the lateral walls of the velopharynx [15].

Positional therapy was known in the past as placing bulky masses on the back of patients, also known as the "tennis ball technique" to prevent supine sleep [16]. A new form of positional therapy is the sleep position trainer (SPT) and can be indicated for patients with positional OSA, defined as a supine AHI that is at least twice as high as compared to the AHI in other positions. SPT is a small, lightweight device that the patient can wear around the chest or neck using a strap during the night. A three-dimensional digital accelerometer is used to measure the sleep position of the patient. When the patient is laying on the back, the device responds with a vibration stimulus to initiate body movement. The device stimulates with a gradually increasing strength and stimulus duration, until a non-supine position is detected. The aim is to make the patient switch positions without full awareness and without waking the patient [16,17]. SPT was found to effectively diminish the percentage of supine sleep, reduce the overall AHI, and improve subjective sleepiness in patients with position-dependent OSA [18].

Palatal surgery is a surgical treatment option for OSA patients that has known different techniques over the last couple of years. Barbed reposition pharyngoplasty (BRP) was developed in 2015 and shows promising results in well-selected patients. It is a simple and secure procedure that can be used as a standalone therapy or in combination with another therapy such as MAD. In brief, the method entails that the posterior pillars are displaced in a more lateral and anterior position to enlarge the oropharyngeal inlet as well as the retropalatal space. Then, the posterior pillar is suspended to the pterygomandibular raphe [19,20]. Expansion sphincter pharyngoplasty (ESP) is almost as efficient as BRP, but it comes with a higher risk of complications [20]. The results of ESP are better when combined with other techniques. The procedure always starts with a bilateral tonsillectomy, followed by identifying and isolating the palatopharyngeal muscle and creating a palatopharyngeal muscle rotation flap [20,21].

Surgical treatment of the upper airway is common for OSA. Hypoglossal nerve stimulation (HNS) or upper airway stimulation is an innovative therapy for patients with moderate to severe OSA. A surgically implanted device will generate respiration synchronized electrical pulses through a generator that is implanted in the upper right chest. These electrical pulses are sent to the hypoglossal nerve to stimulate tongue protrusion and widening of the pharyngeal wall to alleviate upper airway collapse [22,23]. The device consists of a pulse generator, which is implanted just below the right clavicula, and two leads. The sensing lead will be implanted in the second intercostal space close to the right lung to detect breathing. The other lead contains a cuff which will be placed around the protruding branches of the hypoglossal nerve to guide pulses through the nerve and to generate muscle contraction [24]. Postoperatively, the device can be activated at night with a remote after one month. Variable electrode configurations can be installed to obtain an optimal result. The device will be set up during a sleep study one month to six weeks after the procedure. The first ideas about the effect of the HNS can then be observed and the configurations can be changed.

Patients are suitable for HNS following these exclusion criteria: a complete concentric collapse of the palate during DISE, an AHI ≥ 65/h, a BMI ≥ 32 kg/m2, and not having tried CPAP and MAD therapy in the past. Also, confounding sleep disorders and ≥15% central apneas need to be excluded.

Combination therapy for the treatment of obstructive sleep apnea (OSA) is occasionally necessary to achieve optimal outcomes, although it applies to a relatively small subset of patients. For some individuals, a single treatment modality may not sufficiently alleviate symptoms or address the multifactorial nature of their airway obstruction. In such cases, a tailored approach that integrates multiple therapies can be beneficial. For example, combining hypoglossal nerve stimulation, which targets neuromuscular control of the upper airway, with sleep position therapy, which mitigates positional airway collapse, can provide synergistic effects [25]. This dual strategy may be particularly effective for patients with complex anatomical or physiological contributors to their OSA, offering improved symptom relief and enhanced adherence compared to monotherapy. By recognizing and addressing the unique needs of this patient group, healthcare providers can deliver more comprehensive and effective treatment plans [26].

In a case where any alternative treatment to CPAP is considered, drug-induced sleep endoscopy (DISE) is often performed. DISE is a clinical standard diagnostic procedure to study the collapse pattern of the upper airway in patients with snoring and/or sleep apnea problems during drug-induced sleep. It allows us to visualize the upper airway using sedative drugs, which mimic natural sleep [27]. DISE allows us to identify an OSA patient and the characteristics of the upper airway, as collapse patterns differ from patient to patient. With information obtained from DISE, targeted therapy can be considered which is preferred in current days where personalized medicine is the aim [28].

The primary objective of this study is to establish a real-world database that collects patient data seamlessly within the framework of standard clinical care. By integrating data collection into routine patient management, the investigators aim to capture valuable insights into the effectiveness and patient-reported outcomes of alternative treatments for CPAP intolerance.

By this approach, the investigators seek to bridge the gap between research and clinical practice, facilitating the development of evidence-based guidelines and personalized treatment algorithms for patients with CPAP intolerance. By leveraging real-world data, the investigators can improve the quality of care and ultimately enhance the well-being of individuals affected by OSA.

ELIGIBILITY:
Inclusion Criteria:

* adult patients (age starting from 18 years old)
* moderate to severe OSA (AHI ≥ 15/h)
* CPAP-intolerant or non-compliant
* willing to explore alternative treatment options

Exclusion Criteria:

* patients who are still on CPAP therapy
* pediatric patients
* newly diagnosed patients who have not had CPAP before
* patients with AHI ≥ 65 events/h.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (age starting from 18 years old) with moderate to severe OSA (AHI ≥ 15/h) who have been shown to be CPAP-intolerant or non-compliant and are willing to explore alternative treatment options.
Sampling Method: Non-Probability Sample
Enrollment: 850 (Estimated)
Dates: Start 2025-04-28 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
Apnea-hypopnea index (AHI) as measured by a poly(somno)graphy | From baseline to 3 and 12 months
  The AHI is an index of sleep apnea severity that encompasses the frequency of apneas (cessations in breathing) and hypopneas (reductions in airflow) per hour of sleep.

SECONDARY OUTCOMES:
Reason for CPAP intolerance | At baseline
  Patient that return the CPAP device will be asked about the reason of discontinuating the therapy.
Daytime sleepiness measured by the Epworth Sleepiness Scale (ESS) questionnaire | From baseline to 3 and 12 months
  The ESS questionnaire assesses the probability of falling asleep in various settings and situations in daily life. This questionnaire consists of eight questions which can be scored on a four-point Likert-type scale. The lowest score (zero) suggests that the described incident is absent and the highest score (three) suggests the presence of this event. The summation of the eight items can range from 0 to 24.
Disease-specific quality of life as measured by the Functional Outcomes of Sleep Questionnaire-30 (FOSQ-30) questionnaire | From baseline to 3 and 12 months
  The FOSQ-30 is a disease-specific quality of life questionnaire that determines functional status in adults; measures are designed to assess the impact of disorders of excessive sleepiness on multiple activities of everyday living and the extent to which these abilities are improved by effective treatment.
Degree of snoring measured by the Visual Analogue Scale (VAS) questionnaire | From baseline to 3 and 12 months
  Snoring intensity is evaluated using a 10 cm visual analogue scale (VAS) from 0 to 10: 0 represents no snoring, 1-3 represents minimally annoying, 4-6 represents moderately annoying, 7-9 represents annoying, and 10 represents extremely annoying
DISE-score during baseline DISE | At baseline
  DISE-scores (pattern and degree of collapse at each site of upper airway collapse) will be scored

CONTACTS AND LOCATIONS:
Locations (1):
- Universiteit Antwerpen, Wilrijk, Antwerpen, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Van Daele M, Smolders Y, Van Loo D, Bultynck C, Verbraecken J, Vroegop A, Lapperre T, Op de Beeck S, Dieltjens M, Vanderveken OM. Personalized Treatment for Obstructive Sleep Apnea: Beyond CPAP. Life (Basel). 2024 Aug 13;14(8):1007. doi: 10.3390/life14081007. PMID 39202749